CLINICAL TRIAL: NCT04038853
Title: Use of Vitamin D in Treatment of Non-Alcoholic Fatty Liver Disease Detected by Transient Elastography
Brief Title: Vitamin D in Fatty Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Rijeka (Other)
Collaborators: University of Rijeka (Other); Pliva Hrvatska d.o.o. (Unknown)
Responsible Party: Principal Investigator, Ivana Mikolasevic, Asst. Prof., University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00000000-NAFLD
Record Dates: First submitted 2019-07-22; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Non-alcoholic Fatty Liver Disease; Vitamin D Deficiency
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Vitamin D Deficiency | interventions — 1,25-dihydroxyvitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental): Intervention drug, containing 1,25-dihydroxy-vitamin D, comes in original packages as vials containing a total amount of 10 ml of clear solution. 5 drops accounting for 1000 IU of 1,25-dihydroxy-vitamin D will be administered orally on a daily basis.
  Interventions: Drug: 1,25-Dihydroxyvitamin D
- Placebo (Placebo Comparator): A placebo identical to the study intervention drug in all its characteristics (package, visual characteristics of the fluid, smell, and taste) will be administered in the same manner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1,25-Dihydroxyvitamin D — 1,25-dihydroxy-vitamin D3 1000 IU orally daily for 12 months
  Other Names: 1,25-Dihydroxy-Cholecalciferol, Cholecalciferol, Vitamin D3
  Arms: Vitamin D
Drug: Placebo — Placebo identical to the study intervention drug
  Arms: Placebo

SUMMARY:
This study evaluates the influence of vitamin D in reducing laboratory, elastographic (Fibroscan) and metabolic components of NAFLD. Half of the patients will receive vitamin D (Plivit D3) while the other half will receive placebo

DETAILED DESCRIPTION:
In this study will participate patients who come to the regular ambulatory examinations (referred by gastroenterologists, or family physicians in the Department of Gastroenterology CHC Rijeka) and have one or more components of the metabolic syndrome (hypertension, diabetes, obesity, dyslipidemia).Nonalcoholic fatty liver disease will be defined by transient elastography (FibroScan, Echosens, Paris); Controlled Attenuation Parameter (CAP) for assesment of liver steatosis and Liver Stiffness Measurements (LSM) for liver fibrosis. In all patients other causes of chronic liver disease will be excluded; chronic viral hepatitis, autoimmune diseases and other metabolic liver diseases as well as use of drugs than can cause liver steatosis and fibrosis and alcoholic liver disease.

This study will include 450 patients. Taking into account the possible drop-out rate around 15% of the patients during the study period, a total of 400 patients will be randomized. Patients will be randomized into two groups. The first group will be consisted of the patients with NAFLD who will be receiving original medication during the 12 month period. The second group will be consisted of the patients with NAFLD who will be receiving placebo during the 12 months period, which will be identical to the original medication in its packaging and form.

After the 6 and 12 months of therapy in all patients will be evaluated: liver enzymes and metabolic laboratory parameters of NAFLD (insulin resistance, lipidogram and serum glucose), as well as the TE-CAP in order to evaluate the efficiency of Plivit D3 for the treatment of NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* patients with Non-Alcoholic Fatty Liver Disease (NAFLD)
* signed informed consent
* possibility to follow instruction and the protocol

Exclusion Criteria:

* chronic B or C hepatitis
* usage of hepatotoxic drugs in the period of 6 months before inclusion
* chronic kidney insufficiency (grade 4 and 5), hemodialysis
* any other chronic liver disease
* opioid dependancy
* any malignancy
* HIV seropositivity
* alcohol abuse
* pregnancy
* inability to follow the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Elastographic parameter of steatosis | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change of elastographic parameter of steatosis (Controlled Attenuation Parameter; CAP) during the 6 and 12 months period
Elastographic parameter of fibrosis | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change of elastographic parameter of fibrosis (liver stiffness measurements; LSM) during the 6 and 12 months period

SECONDARY OUTCOMES:
Aspartate transaminase | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change in liver enzyme aspartate transaminase (AST) serum levels in the period of 6 and 12 months. Normal range = 11-38 IU/L.
Alanine transaminase | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change in liver enzyme alanine transaminase (ALT) serum levels in the period of 6 and 12 months. Normal range = 12-48 IU/L.
Gamma-glutamyl transferase | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change in liver enzyme gamma-glutamyl transferase (GGT) serum levels in the period of 6 and 12 months. Normal range = 11-55 IU/L.
Insuline Resistance | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change in insulin resistance defined by the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR; normal range = 0.5 to 1.4) score in the period of 6 and 12 months
Total cholesterol | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change in total cholesterol serum levels in the period of 6 and 12 months
Low-density lipoprotein | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change in low-density lipoprotein (LDL) serum levels in the period of 6 and 12 months
High-density lipoprotein | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change in high-density lipoprotein (HDL) serum levels in the period of 6 and 12 months
Triglyceride | Week 0 - initiation; after 6 months; and after 12 months (end of study)
  Change in triglyceride (TG) serum levels in the period of 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Mikolasevic, MD, PhD, Principal Investigator — Department of Gastroenterology, Clinical Hospital Center Rijeka, University of Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No